CLINICAL TRIAL: NCT05855395
Title: A Bidimensional Early Intervention Strategy of Standard of Care Combined With Host Immunomodulation in Elderly Patients With Mild or Moderate COVID-19: A Multicentre, Randomized, Controlled, Adaptive Platform Study
Brief Title: The Standard of Care Combined With Glucocorticoid in Elderly People With Mild or Moderate COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases Affiliation: Huashan Hospital, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEAT-COV
Record Dates: First submitted 2023-02-27; First posted 2023-05-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: Glucocorticoids; Standard of care; Mild and moderate COVID-19
MeSH Terms: conditions — COVID-19; Lymphoma, Follicular | interventions — Glucocorticoids; Dexamethasone; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Experimental group with standard of care combined with glucocorticoid（dexamethasone: 3mg qd x 5 days; or prednisone: 20mg qd x 5 days; or methylprednisolone: 16mg qd x 5 days)
  Interventions: Drug: Glucocorticoid
- Group B (No Intervention): Control group with standard of care（The clinical standard of care of COVID-19 includes general treatment, oral antiviral drugs, immunotherapy, oxygen therapy and respiratory support, etc.）

INTERVENTIONS:
Drug: Glucocorticoid — standard of care combined with glucocorticoid(dexamethasone: 3mg qd x 5 days; or prednisone: 20mg qd x 5 days; or methylprednisolone: 16mg qd x 5 days)
  Other Names: dexamethasone; prednisone; methylprednisolone
  Arms: Group A

SUMMARY:
This study is aimed to explore the dual-dimensional early intervention strategy of standard of care combined with host immunomodulation in elderly patients with mild and moderate COVID-19.

DETAILED DESCRIPTION:
In this multicentre, randomized, controlled, and adaptive platform trial exploring the efficacy and safety of short-term and low-dose glucocorticoid combined with standard of care in mild or moderate elderly patients (with or without other high-risk factors) who are over 65 years.We are looking for the best treatment strategy to prevent mild or moderate COVID-19 from developing into severe/critical COVID-19, so as to reduce the risk of disease progression and death in the elderly patients and benefit more patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65;
* Male or female;
* Positive test for coronavirus antigen or nucleic acid；
* Within 7 days of onset (fever and/or cough) ；
* mild and moderate；Mild: respiratory tract infection is the main manifestation, such as dry throat, sore throat, cough, fever；Moderate: continuous high fever>3 days or (and) cough, shortness of breath, etc., but respiratory rate (RR)<30 times/minute, oxygen saturation>93% when breathing air at rest. Imaging findings of characteristic pneumonia caused by COVID-19 infection；
* The patient is willing to participate in the trial treatment and follow-up, and sign the informed consent form (if the patient lacks the ability to give informed consent due to his serious medical condition, such as acute respiratory failure or the need for respiratory support, he can obtain the consent of the patient's legal representative)；
* No systemic glucocorticoids treatment in the past 7 days；

Exclusion Criteria:

* Serious and uncontrolled comorbidities；
* Expected lifetime is less than 1 month；
* Severe/critical;
* Other situations that are evaluated by researchers as not suitable for participating the study.

Criteria for discontinuation

* The subject could not benefit after treatment (discontinued patients could be analyzed according to the PP analysis set);

Withdrawal criteria (if any of the following items are required)

* The subject asked to withdraw from the study;
* The subject needs to withdraw from the study after clinical observation after discontinuing treatment;
* The subject died or lost to follow-up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5815 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who progress to severe or critical COVID-19 within 28 days | In 28 days
  Definition of severe COVID-19
  1. At rest, oxygen saturation ≤ 93% when inhaling air;
  2. Progression due to COVID-19 (defined as >50% of significant progression of lesions within 24~48 hours on lung imaging; or respiratory failure requiring mechanical ventilation; or emergency department visits or hospitalizations with shock) and/or complications (comitant other organ failure requiring intensive care unit monitoring).

SECONDARY OUTCOMES:
Duration of antigen or nucleic acid negative conversion | In 28 days
  Duration of antigen or nucleic acid negative conversion
Day 14 antigen or nucleic acid conversion rate | Day 14
  Day 14 antigen or nucleic acid conversion rate
Time for initial symptom relief，Duration of symptom relief | In 14 days
  Time for initial all symptoms relief (Date when symptoms were first reported as mild or asymptomatic), Duration of all symptoms relief(The date when all symptoms were first reported as mild or asymptomatic, followed by remaining mild or asymptomatic until the 14th day）
All-cause mortality | In 28 days
  Short-term case fatality rate defined in the study, including case fatality on day 28
Days of respiratory symptoms | In 28 days
  Days of respiratory symptoms
Duration of outpatient hospitalization/emergency department visits due to COVID-19 progression(from the date of enrollment) | In 28 days
  Duration of outpatient hospitalization/emergency department visits due to COVID-19 progression(from the date of enrollment)
Length of hospital stay for any reason | In 28 days
  Length of hospital stay for any reason
Proportion of patients who progress to severe or critical COVID-19 within 28 days | In 28 days
  Oxygen saturation ≤ 93% when inhaling air at rest
Proportion of emergency department visits or hospitalizations due to COVID-19 progression | In 28 days
  Progression due to COVID-19 (defined as >50% of significant progression of lesions within 24~48 hours on lung imaging; or respiratory failure requiring mechanical ventilation; or emergency department visits or hospitalizations with shock) and/or complications (comitant other organ failure requiring intensive care unit monitoring).

OTHER OUTCOMES:
ADRs and SADRs associated with glucocorticoid therapy and antiviral therapy（One of the standard treatments) were collected | In 14 days
  ADRs and SADRs associated with glucocorticoid therapy and antiviral therapy（One of the standard treatments) were collected

CONTACTS AND LOCATIONS:
Overall Officials: WenHong Zhang, M.D., Principal Investigator — Huashan Hospital
Locations (15):
- China (15):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Quanzhou First Hospital, Quanzhou, Fujian
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Attached Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Huaihua First People's Hospital, Huaihua, Hunan
  - Nanjing Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Wuxi Fifth People's Hospital, Wuxi, Jiangsu
  - The People's Hospital Of Xingguo County, Ganzhou, Jiangxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - The First People's Hospital Of YunNan, Kunming, Yunnan
  - People's Hospital of Qiubei County, Yunnan Province, Wenshan, Yunnan
  - Hangzhou Linping District First People's Hospital, Hanzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
After thesis defense the study will be published internationally to be available for the public.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within two year
Access Criteria: Not yet

REFERENCES:
- [Background] Agusti A, De Stefano G, Levi A, Munoz X, Romero-Mesones C, Sibila O, Lopez-Giraldo A, Plaza Moral V, Curto E, Echazarreta AL, Marquez SE, Pascual-Guardia S, Santos S, Marin A, Valdes L, Saldarini F, Salgado C, Casanovas G, Varea S, Rios J, Faner R. Add-on inhaled budesonide in the treatment of hospitalised patients with COVID-19: a randomised clinical trial. Eur Respir J. 2022 Mar 10;59(3):2103036. doi: 10.1183/13993003.03036-2021. Print 2022 Mar. PMID 35144989
- [Background] Song JY, Yoon JG, Seo YB, Lee J, Eom JS, Lee JS, Choi WS, Lee EY, Choi YA, Hyun HJ, Seong H, Noh JY, Cheong HJ, Kim WJ. Ciclesonide Inhaler Treatment for Mild-to-Moderate COVID-19: A Randomized, Open-Label, Phase 2 Trial. J Clin Med. 2021 Aug 12;10(16):3545. doi: 10.3390/jcm10163545. PMID 34441840
- [Background] Agarwal A, Hunt B, Stegemann M, Rochwerg B, Lamontagne F, Siemieniuk RA, Agoritsas T, Askie L, Lytvyn L, Leo YS, Macdonald H, Zeng L, Alhadyan A, Muna A, Amin W, da Silva ARA, Aryal D, Barragan FAJ, Bausch FJ, Burhan E, Calfee CS, Cecconi M, Chacko B, Chanda D, Dat VQ, De Sutter A, Du B, Freedman S, Geduld H, Gee P, Haider M, Gotte M, Harley N, Hashimi M, Hui D, Ismail M, Jehan F, Kabra SK, Kanda S, Kim YJ, Kissoon N, Krishna S, Kuppalli K, Kwizera A, Lado Castro-Rial M, Lisboa T, Lodha R, Mahaka I, Manai H, Mendelson M, Migliori GB, Mino G, Nsutebu E, Peter J, Preller J, Pshenichnaya N, Qadir N, Ranganathan SS, Relan P, Rylance J, Sabzwari S, Sarin R, Shankar-Hari M, Sharland M, Shen Y, Souza JP, Swanstrom R, Tshokey T, Ugarte S, Uyeki T, Evangelina VC, Venkatapuram S, Vuyiseka D, Wijewickrama A, Tran L, Zeraatkar D, Bartoszko JJ, Ge L, Brignardello-Petersen R, Owen A, Guyatt G, Diaz J, Kawano-Dourado L, Jacobs M, Vandvik PO. A living WHO guideline on drugs for covid-19. BMJ. 2020 Sep 4;370:m3379. doi: 10.1136/bmj.m3379. PMID 32887691
- [Background] Orchard K, Dignan FL, Lee J, Pearce R, Desai M, McFarlane E, Parkin A, Shearn P, Snowden JA. The NICE COVID-19 rapid guideline on haematopoietic stem cell transplantation: development, implementation and impact. Br J Haematol. 2021 Feb;192(3):467-473. doi: 10.1111/bjh.17280. Epub 2021 Jan 20. No abstract available. PMID 33474730
- See also: Guide：Diagnosis and Treatment Plan for COVID-19 (Tenth Edition on Trial) — http://www.gov.cn/xinwen/2023-01/06/content_5735357.htm